CLINICAL TRIAL: NCT02583438
Title: Beijing Chao-yang Hospital, Capital Medical University
Brief Title: Evaluate the Effect of Saxagliptin on Gut Microbiota in Patients With Newly Diagnosed Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Department of Endocrinology, Beijing Chao Yang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Saxa015
Record Dates: First submitted 2015-10-14; First posted 2015-10-22 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Gut Microbiota; inflammatory marker; Glucose and lipid metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle intervention (Experimental)
  Interventions: Drug: Saxagliptin (Bristol-Myers Squibb Company)

INTERVENTIONS:
Drug: Saxagliptin (Bristol-Myers Squibb Company) — 6-month treatment of Saxagliptin 5mg Qd

SUMMARY:
The intestinal microflora imbalance has been associated with obesity and type 2 diabetes. The researchers' study aimed to investigate the effect of saxagliptin on gut microbiota in patients with newly diagnosed type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Females or males, and aged 20 to 65 years.
* Newly diagnosed type 2 diabetes
* HbA1C ≥7% and HbA1C <9%

Exclusion Criteria:

* Hepatic insufficiency (ALT or AST> 1.5*ULN)
* Renal insufficiency [Creatinine clearance rate (Ccr)]<60ml/min estimated from MDRD equation)
* Coronary artery disease
* Thyroid disease
* Infectious disease
* Systemic inflammatory disease
* Cancer
* Subjects who were taking agents known to influence gut microbiota
* Pregnant or lactating woman
* Other conditions at investigator's discretion

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
gut microbiota | Change from Baseline Bacteroidetes abundances and composition of gut microbiota at 6 months

SECONDARY OUTCOMES:
The improvement of intestinal microflora imbalance | Bacteroidetes abundances and composition of gut microbiota (baseline, 4 weeks, 8 weeks and 12 weeks)
The change of inflammatory markers | The change of inflammatory markers (baseline, 12 weeks)
  The effect on plasma levels of inflammatory markers, such as IL-1B, IL-6 and TNF-α(baseline, 12 weeks)